CLINICAL TRIAL: NCT06038227
Title: Comparing Outcomes for Minimally Invasive Techniques for Anatomic Lung Resection for Cancer - A Prospective, Comparative, Non-randomized, Open Label Post-market Observational Cohort Study Within Europe
Brief Title: Lung cAncer Robotic Comparative Study
Acronym: LARCS
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1114332C
Record Dates: First submitted 2023-08-24; First posted 2023-09-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
Keywords: Minimally invasive surgery; Robotics
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Robotic Assisted Thoracic Surgery: Participants will undergo robotic assisted thoracic surgery (RATS) for segmentectomy or lobectomy.
  Interventions: Procedure: Robotic Assisted Thoracic Surgery
- Video Assisted Thoracic Surgery: Participants will undergo video assisted thoracic surgery (VATS) for segmentectomy or lobectomy.
  Interventions: Procedure: Video Assisted Thoracic Surgery

INTERVENTIONS:
Procedure: Robotic Assisted Thoracic Surgery — Surgeons will pre-determine to perform a segmentectomy or lobectomy using RATS.
  Groups: Robotic Assisted Thoracic Surgery
Procedure: Video Assisted Thoracic Surgery — Surgeons will pre-determine to perform a segmentectomy or lobectomy using VATS.
  Groups: Video Assisted Thoracic Surgery

SUMMARY:
To compare outcomes of minimally invasive surgical techniques for the treatment of early-stage non-small cell lung cancer.

DETAILED DESCRIPTION:
Detection of lung cancer is occurring at increasingly earlier stages due to improved screening and the discovery of incidental nodules. Coinciding with this trend is recent data from two international randomized, control trials, RAVAL - (Robotic Lobectomy vs. Thoracoscopic Lobectomy for Early Stage Lung Cancer) and, JCOG0802 (The Japan Clinical Oncology Group) that show oncologic outcomes from segmentectomy are equivalent to lobectomy for cancers ≤2 cm. However, segmentectomy is a more complex technical operation that may not be easily feasible using video assisted thoracic surgery (VATS) but could be facilitated by robotic-assisted thoracic surgery (RATS), allowing improved vision, precision and controlled anatomic dissection.

The LARCS study is designed to understand the perioperative outcomes of patients and identify the real-world selection process of either VATS and RATS segmentectomy and lobectomy for lung cancers ≤2 cm. It aims to generate evidence to support integration of patient-centered care using minimally invasive technology.

In addition, health related quality of life captured in the study will also provide valuable insight into time to recovery, determining burden of the disease, and guide future treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with clinical stage IA1-2 non-small cell lung cancer at time of procedure
* Patient scheduled to undergo minimally invasive surgery for NSCLC with either da Vinci robotic assisted surgery or VATs
* Aged ≥ 18 years
* Must be willing and able to comply with study requirements
* Must indicate their understanding of the study and willingness to participate by signing an appropriate informed consent form

Exclusion Criteria:

* Patients with clinical stage IA3, II, III, and IV lung cancer
* Patient receiving a lobectomy/segmentectomy as an emergency procedure
* Patients receiving a lobectomy/segmentectomy for metastatic cancer
* Patients scheduled to receive a bilobectomy or sleeve-lobectomy
* Mental incapacity to understand or consent to study procedures
* Anticipated difficulty for patient to comply with protocol requirements
* Unable to comply with the follow up schedule
* Pregnant or are planning to become pregnant during the study
* Life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from adult participants who have a lobectomy or segmentectomy for treatment of non small cell lung cancer (clinical stages IA1-2) will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient reported Quality of Life 1 | 1 month post surgery
  EQ 5D 5L (European Quality of Life Five Dimension) The EQ-5D-5L is a validated and established generic Patient Reported Outcome (PRO) instrument that uses 6 questions to assess patients' quality of life. It includes a vertical EQ visual analog scale (EQ VAS, 0-100 points) and a descriptive EQ-5D-5L system. An algorithm is used to calculate the scores.
  For the descriptive section of the scale, an index value of 1 represents the best possible health state, while an index value of <0 (variable) represents the worst possible health state.
  The EQ VAS score is rated on a scale of 0-100 points. 0 points correspond to the worst possible health status, while 100 points correspond to the best possible health status.
Patient reported Quality of Life 2 | 1 month post surgery
  RNLI (Reintegration to Normal Living Index) The RNLI has 11 questions and is scored on a visual analogue scale (VAS). On one end: "does not describe my situation" (1 or minimal integration) and "fully describes my situation" (10 or complete integration). Individual item scores are summed to provide the total score. The higher the score, the better the patients perceived integration.

SECONDARY OUTCOMES:
Number of conversions from pre-operative surgical plan | immediately post operative
  Number of participants who undergo conversion surgery from the pre-operative surgical plan captured on the surgical decision making form. Conversion may be from segmentectomy to lobetomy, RATS or VATS to open surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Routledge, Principal Investigator — Guy's St Thomas' NHS Foundation Trust, UK; Rune Eggum, Principal Investigator — University Hospital, Akershus; Martin Eichhorn, Principal Investigator — Thoraxklinik Heidelberg, Germany
Locations (11):
- France (3):
  - AP-HM, Marseille
  - CHU de Rouen, Rouen
  - CHU de Toulouse, Toulouse
- Germany (2):
  - Thoraxklinik, Heidelberg
  - Krankenhaus Barmherzige Brüder, Regensburg
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy
- Akershus University Hospital, Loerenskog, Norway
- United Kingdom (4):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Guy's and St Thomas' NHS Foundation Trust, London
  - St Bartholomew Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel YS, Hanna WC, Fahim C, Shargall Y, Waddell TK, Yasufuku K, Machuca TN, Pipkin M, Baste JM, Xie F, Shiwcharan A, Foster G, Thabane L. RAVAL trial: Protocol of an international, multi-centered, blinded, randomized controlled trial comparing robotic-assisted versus video-assisted lobectomy for early-stage lung cancer. PLoS One. 2022 Feb 2;17(2):e0261767. doi: 10.1371/journal.pone.0261767. eCollection 2022. PMID 35108265
- [Background] Saji H, Okada M, Tsuboi M, Nakajima R, Suzuki K, Aokage K, Aoki T, Okami J, Yoshino I, Ito H, Okumura N, Yamaguchi M, Ikeda N, Wakabayashi M, Nakamura K, Fukuda H, Nakamura S, Mitsudomi T, Watanabe SI, Asamura H; West Japan Oncology Group and Japan Clinical Oncology Group. Segmentectomy versus lobectomy in small-sized peripheral non-small-cell lung cancer (JCOG0802/WJOG4607L): a multicentre, open-label, phase 3, randomised, controlled, non-inferiority trial. Lancet. 2022 Apr 23;399(10335):1607-1617. doi: 10.1016/S0140-6736(21)02333-3. PMID 35461558
- See also: Protocol of an international, multi-centered, blinded, randomized controlled trial comparing robotic-assisted versus video-assisted lobectomy for early-stage lung cancer — https://pubmed.ncbi.nlm.nih.gov/35108265/
- See also: Segmentectomy versus lobectomy in small-sized peripheral non-small-cell lung cancer (JCOG0802/WJOG4607L): a multicentre, open-label, phase 3, randomised, controlled, non-inferiority trial. — https://pubmed.ncbi.nlm.nih.gov/35461558/